CLINICAL TRIAL: NCT05730985
Title: Effectiveness of the Intake of a Food Supplement Based on Hydroxymethylbutyrate, Carnosine, Lactoferrin and Magnesium on Reduction of Inflammation and on the Improvement of the Health of the Muscle
Brief Title: From the Gut to the Strut: Reducing Inflammation for Healthy Muscles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1206/01072022
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Inflammation; Sarcopenia; Gut Permeability
MeSH Terms: conditions — Inflammation; Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intevention group (Experimental): Experimental formula (Miotrof®) to take 1 sachet per day for 4 months
  Interventions: Dietary Supplement: Miotrof® formula
- Placebo group (Placebo Comparator): Placebo formula to take 1 sachet per day for 4 months
  Interventions: Dietary Supplement: Placebo formula

INTERVENTIONS:
Dietary Supplement: Miotrof® formula — 1 sachet per day for 4 months
  Arms: Intevention group
Dietary Supplement: Placebo formula — 1 sachet per day for 4 months
  Arms: Placebo group

SUMMARY:
This research aims to evaluate the effectiveness of a dietary supplement on reducing inflammation and improving muscle health. The product is a food supplement notified to the Ministry of Health consisting of: hydroxymethylbutyrate, carnosine, lactoferrin and magnesium, which help reduce inflammation and intestinal permeability and to improve muscle health.

ELIGIBILITY:
Inclusion Criteria:

* sarcopenic patients aged 55-85. Sarcopenia will be diagnosed according to the European Working Group on Sarcopenia in Older People (EWSGOP-2) criteria by muscle strength or chair stand test.

Exclusion Criteria:

* severe kidney disease (glomerular filtration rate <30 mL/min),
* moderate-to-severe hepatic failure (Child-Pugh Class of B or C),
* endocrine diseases associated with disorders of calcium metabolism (with the exception of osteoporosis),
* psychiatric disorders,
* cancer (in the previous 5 years),
* hypersensitivity to any investigational food component
* subjects taking protein/amino acid supplements (up to 3 months prior to the study).
* patients not capable of taking oral therapy and those receiving or having indication for artificial nutrition or included in another clinical nutrition trial

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Inflammation status | At the beginning of the treatment
  A blood sample will be collected and analised for C-reactive protein and tumor necrosis factor alfa (TNF alfa)
Inflammation status | After 4 months of treatment
  A blood sample will be collected and analised for C-reactive protein and tumor necrosis factor alfa (TNF alfa)
Muscle strength evaluation | At the beginning of the treatment
  Muscle strength was measured by handgrip strength according to standard procedures by a hydraulic hand dynamometer (Jamar 5030 J1, Sammons Preston Rolyan, Bolingbrook, Canada with an accuracy of 0.6 N). The subject holds the dy-namometer in the hand to be tested, with the arm at right angles and the elbow by the side of the body, applying an isometric contraction
Muscle strength evaluation | After 4 months of treatment
  Muscle strength was measured by handgrip strength according to standard procedures by a hydraulic hand dynamometer (Jamar 5030 J1, Sammons Preston Rolyan, Bolingbrook, Canada with an accuracy of 0.6 N). The subject holds the dy-namometer in the hand to be tested, with the arm at right angles and the elbow by the side of the body, applying an isometric contraction
body composition assessment | At the beginning of the treatment
  Body composition represented by fat free mass and fat mass were measured using a Lunar Prodigy DXA (GE Medical Systems, WI, USA).
body composition assessment | After 4 months of treatment
  Body composition represented by fat free mass and fat mass were measured using a Lunar Prodigy DXA (GE Medical Systems, WI, USA).
Physical performance assessment | At the beginning of the treatment
  Physical performance was assessed using the Short Physical Performance battery test (SPPB) which comprised of gait speed, chair-stand test, and balance (three different tests that assess the ability to stand with the feet together in the side-by-side, semi-tandem, and tandem positions); each component was scored from 0 (not possible) to 4 (best performance) and the scores were added up to a total score ranging from 0 to 12.
Physical performance assessment | After 4 months of treatment
  Physical performance was assessed using the Short Physical Performance battery test (SPPB) which comprised of gait speed, chair-stand test, and balance (three different tests that assess the ability to stand with the feet together in the side-by-side, semi-tandem, and tandem positions); each component was scored from 0 (not possible) to 4 (best performance) and the scores were added up to a total score ranging from 0 to 12.
Gut permeability. | At the beginning of the treatment
  A blood sample will be collected and analised for indican
Gut permeability. | After 4 months of treatment
  A blood sample will be collected and analised for indican

CONTACTS AND LOCATIONS:
Locations (1):
- l'Istituto di Riabilitazione e cura "Santa Margherita" di Pavia, Azienda di Servizi alla Persona (ASP)., Pavia, Italy